CLINICAL TRIAL: NCT00668616
Title: Cyclophosphamid + Farmorubicin® With Subsequent Administration of Taxol® (q3w) Versus Intensified Administration of Farmorubicin® Followed by Taxol® (q2w) in the Adjuvant Treatment of Breast Cancer in Patients With 1-3 Afflicted Lymph Nodes (1-3 LK+)
Brief Title: Adjuvant Treatment of Breast Cancer With 1-3 Aflicted Lymph Nodes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170200
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer
Keywords: breast cancer with 1-3 afflicted axillary lymph nodes
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Paclitaxel; Filgrastim

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Cyclophosphamide, Epirubicin, Paclitaxel
- 2 (Experimental)
  Interventions: Drug: Epirubicin, Paclitaxel, Filgrastim

INTERVENTIONS:
Drug: Cyclophosphamide, Epirubicin, Paclitaxel — 4 cycles of 600 mg/m² cyclophosphamide i.v. and 90 mg/m2 Farmorubicin i.v. on day 1, q21d followed by 4 cycles of 175 mg/m² Taxol, day 1, q21d
  Arms: 1
Drug: Epirubicin, Paclitaxel, Filgrastim — cycle 1-4: 120 mg/m² Epirubicin i.v. on day 1, q14d, 5 µg/kg s.c. filgrastim day 5-10 (if leucocytes are lower than 10000/µl) cycle 5-8: 175 mg/m² Paclitaxel i.v. on day 1, q14d, 5 µg/kg s.c. filgrastim day 5-10 (if leucocytes are lower than 10000/µl)
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether a treatment with 4 cycles anthracycline + cyclophoshamide followed by administration of 4 cycles paclitaxel is more effective than therapy with 4 cy<cles of anthracycline adminbistration followed by 4 cycles of paclitaxel

ELIGIBILITY:
Inclusion Criteria:

* women with histologically proven breast cancer (pT1/pT2/pT3, pN1, N0)
* ECOG performance status 0-1
* start of adjuvant therapy not later than 4 weeks after surgery
* hematology: platelets at least 100xGpt/l, neutrophiles at least 2xGpt/l
* normal liver function as defined by: bilirubine till 1.5 x normal value, SGOT/SGPT till 1.25 x normal value
* normal kidney function as defined by: creatine till 1.5 x normal value
* negative pregnancy test for patients before menopause and effective contraception
* written informed consent

Exclusion Criteria:

* prior radiation, chemotherapy, hormontherapy and immunotherapy
* patients with more than 3 afflicted lymph nodes
* afflicted lymph nodes on the cantralateal side and/or afflicted supraclavicular or intraclavicular lymph nodes
* bilateral breast cancer or second carcinoma of the breast
* inflammatory breast cancer and/or distant metastases
* existing clinically relevant peripheral neuropathie
* heart infection during the last 6 months or therapeutically not compensated heart failure or cardiac arrhythmias of at least LOWN II
* patients with active infections and/or not controlled hypercalcemia
* pregnant or breastfeeding women or women of child-bearing age who do not use effictive contrazeptiva

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1034 (Actual)
Dates: Start 2000-03; Primary Completion 2005-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
progression-free time | every 3-6 months

SECONDARY OUTCOMES:
toxicity
overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Oskar-Ziethen-Krankenhaus, Berlin, State of Berlin, Germany